CLINICAL TRIAL: NCT05928689
Title: Misophonia-Related Memory Modification Using Reconsolidation Mechanisms: Pharmacological and Behavioral Manipulation
Brief Title: Behavioral and Pharmacological Reconsolidation Interference in Misophonia
Acronym: Miso Prop
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniela Schiller, Professor of Neuroscience and Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY-22-01280
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Misophonia
MeSH Terms: conditions — misophonia | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: The study team will measure reactivity to misophonia-related cues following either a pharmacological manipulation via a 40 mg propranolol tablet or behavioral manipulation via counterconditioning.
  The study team predicts that participants with misophonia who experience a reminder (reactive a misophonia memory) and receive the pharmacological or behavioral manipulation, will show reduced reactivity to misophonia cues.
  Other groups that undergo one of these components alone (reminder only, drug only, counterconditioning only) will continue to show heightened reactivity to misophonia cues.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is multi-arm and single-site randomized study that is placebo-controlled and single- and double-blinded depending on the condition assignment. Some groups will experience reminders, or short exposures to misophonia-related cues. Some groups will take the study intervention, propranolol hydrochloride (or matching placebo) oral tablets, and some will undergo counterconditioning, by presenting the misophonia cues with monetary rewards (in a continuous reinforcement schedule with fixed monetary amounts).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Memory Reminder followed by Propranolol Hydrochloride (Experimental): This arm aims to have 30 participants with a pharmacological manipulation. They will receive a reminder to reactivate their memory of a misophonia trigger followed by ingestion of a propranolol hydrochloride tablet.
  Interventions: Drug: Propranolol Hydrochloride tablet; Behavioral: Reminder
- Memory reminder followed by Placebo (Placebo Comparator): This arm aims to have 30 participants with a pharmacological manipulation. They will receive a reminder to reactivate their memory of a misophonia trigger followed by ingestion of a placebo tablet.
  Interventions: Behavioral: Reminder; Drug: Placebo
- No memory reminder followed by Propranolol Hydrochloride (Experimental): This arm aims to have 30 participants with a pharmacological manipulation. They will not receive a reminder to reactivate their memory of a misophonia sound and only receive a propranolol hydrochloride tablet.
  Interventions: Drug: Propranolol Hydrochloride tablet
- Memory reminder followed by counterconditioning (Experimental): This arm aims to have 30 participants with a behavioral manipulation. They will receive a reminder to reactivate their memory of a misophonia trigger and then will undergo counterconditioning.
  Interventions: Behavioral: Reminder; Behavioral: Counterconditioning
- No memory reminder followed by counterconditioning (Experimental): This arm aims to have 30 participants with a behavioral manipulation. They will not receive a reminder to reactivate their memory of a misophonia trigger and then undergo counterconditioning.
  Interventions: Behavioral: Counterconditioning

INTERVENTIONS:
Drug: Propranolol Hydrochloride tablet — Single dose of 40 mg propranolol tablet
  Arms: Memory Reminder followed by Propranolol Hydrochloride; No memory reminder followed by Propranolol Hydrochloride
Behavioral: Reminder — Reactivation of misophonia trigger memory
  Arms: Memory Reminder followed by Propranolol Hydrochloride; Memory reminder followed by Placebo; Memory reminder followed by counterconditioning
Behavioral: Counterconditioning — Counterconditioning will consist of presentation of misophonia cues paired with monetary rewards.
  Arms: Memory reminder followed by counterconditioning; No memory reminder followed by counterconditioning
Drug: Placebo — Matching placebo tablet
  Arms: Memory reminder followed by Placebo

SUMMARY:
One of the core processes presumably underlying misophonia - a condition characterized by decreased tolerance for specific sounds - is associative learning. Using behavioral, computational, and neural analyses of emotional learning and memory processes to understand the unknown behavioral and neural mechanisms underlying misophonia's associative learning and memory, the study team will evaluate whether interference with the reconsolidation of a reactivated misophonia memory with propranolol can alleviate aversive reaction to misophonia-related cues.

ELIGIBILITY:
Inclusion Criteria:

* Hypersensitive to presence of a specific sound, which may be accompanied by irritation, anger/outbursts, or fear.
* Must be between the ages of 18 - 55.
* Must be fluent in English since the study's instructions, surveys, and tasks will be in English

Exclusion Criteria:

* Disability or medical condition that prohibits completion of study. Participants must be able to complete all study procedures to ensure optimal conditions for data analysis.
* CNS disease, such as history of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), or other neurological disease, history of head trauma (defined as loss of consciousness>3 min), or history of seizures without a resolved etiology. CNS disease and drugs that act in the peripheral or central nervous system are likely to have effects on patterns of neural activity. We wish to minimize confounding variables.
* Recently used drugs of abuse.
* Pregnancy. The risks associated with neither propranolol exposure during gestation have been studied extensively. We wish to safeguard the health of potential participants and their children.
* Lactation. Propranolol is excreted in human breast-milk, and its impact on infant development has not been studied. We wish to safeguard the health of potential participants and their children.
* Regular use of medication metabolized in the CYP2D6, 1A2, or 2C19 pathways. Drugs that are metabolized in the same pathway as propranolol may increase its efficacy or toxicity. We wish to safeguard the health of participants.
* Blood pressure over 150/100 or under 100/60 (applicable for either systolic or diastolic measures) and any hypertension requiring medication. Propranolol is known to pose additional risk to individuals with a number of medical conditions. We wish to safeguard the health of our participants.
* Pulse over 100 or under 55.
* History of cardiovascular illness such as cardiac arrhythmia, coronary heart disease or any cardiac dysfunction that requires medication.
* Active respiratory illness including bronchospastic pulmonary disease and chronic obstructive pulmonary disease
* Diabetes mellitus.
* Other medical conditions that make it unsafe to take propranolol (e. g. allergy to propranolol).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in average Galvanic skin response based on deflections of a wave | Baseline and after 6 hours
  Using galvanic skin response based on deflections of a wave, a difference between the average response to the misophonia-related video before and after the pharmacological or behavioral manipulation will be measured. The difference in scores across conditions will be compared. A greater deflection indicates greater sympathetic nervous system arousal.
Change in average heart rate | Baseline and after 6 hours
  Using heart rate measurement, a difference between the average response to the misophonia-related video before and after the pharmacological or behavioral manipulation will be measured. The difference in scores across conditions will be compared. Reduced heart rate will indicate manipulation efficacy
Change in Approach-Avoidance test | Baseline and after 6 hours
  Using an approach-avoidance test, the difference between the monetary amounts earned before and after the pharmacological or behavioral manipulation will be measured. The minimum monetary amount earned is $0 and the maximum monetary amount earned is $23. A higher monetary amount earned indicates greater approach towards an avoidant cue. The difference in monetary amounts across conditions will be compared.

SECONDARY OUTCOMES:
Change in Approach-Avoidance test | about 1 week later
  Using an approach-avoidance test, the difference between the monetary amounts earned before and after the pharmacological or behavioral manipulation will be measured. The minimum monetary amount earned is $0 and the maximum monetary amount earned is $23. A higher monetary amount earned indicates greater approach towards an avoidant cue. The difference in monetary amounts across conditions will be compared.
Change in Approach-Avoidance test | Baseline and 1 month later
  Using an approach-avoidance test, the difference between the monetary amounts earned before and after the pharmacological or behavioral manipulation will be measured. The minimum monetary amount earned is $0 and the maximum monetary amount earned is $23. A higher monetary amount earned indicates greater approach towards an avoidant cue. The difference in monetary amounts across conditions will be compared.
Change in decision making task | Baseline and after 6 hours
  Using a decision making task based on choice behavior (choosing the correct machine more often), the study team will fit computational models to understand reactivity to misophonia-related cues across conditions.
  The study team will measure a difference in the task responses after the pharmacological or behavioral manipulation. Measures will include learning rate, and a link between prediction error and self-reported mood. The scores across conditions will be compared.
Change in decision making task | Baseline and about 1 week
  Using a decision making task based on choice behavior (choosing the correct machine more often), the study team will fit computational models to understand reactivity to misophonia-related cues across conditions.
  The study team will measure a difference in the task responses after the pharmacological or behavioral manipulation. Measures will include learning rate, and a link between prediction error and self-reported mood. The scores across conditions will be compared.
Change in decision making task | Baseline and 1 month later
  Using a decision making task based on choice behavior (choosing the correct machine more often), the study team will fit computational models to understand reactivity to misophonia-related cues across conditions.
  The study team will measure a difference in the task responses after the pharmacological or behavioral manipulation. Measures will include learning rate, and a link between prediction error and self-reported mood. The scores across conditions will be compared.
Change in Average Galvanic skin response based on deflections of a wave | about 1 week later
  Using galvanic skin response based on deflections of a wave, a difference between the average response to the misophonia-related video before and after the pharmacological or behavioral manipulation will be measured. The difference in scores across conditions will be compared. A greater deflection indicates greater sympathetic nervous system arousal.
Change in Average Galvanic skin response based on deflections of a wave | about 1 month later
  Using galvanic skin response based on deflections of a wave, a difference between the average response to the misophonia-related video before and after the pharmacological or behavioral manipulation will be measured. The difference in scores across conditions will be compared. A greater deflection indicates greater sympathetic nervous system arousal.
Change in average heart rate | about 1 week later
  Using heart rate measurement, a difference between the average response to the misophonia-related video before and after the pharmacological or behavioral manipulation will be measured. The difference in scores across conditions will be compared. Reduced heart rate will indicate manipulation efficacy
Change in average heart rate | about 1 month later
  Using heart rate measurement, a difference between the average response to the misophonia-related video before and after the pharmacological or behavioral manipulation will be measured. The difference in scores across conditions will be compared. Reduced heart rate will indicate manipulation efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Schiller, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; James Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Laili Soleimani, MD, Msc, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will publicly share analyzed statistical summaries which are sufficient for data assessment, reanalysis, and meta-analysis, and reproduction of figures.
Time Frame: 2 months after publication
Access Criteria: Open access with no restrictions